CLINICAL TRIAL: NCT02906995
Title: An Open-Label Pseudorandomized, Two Way Crossover Comparison of the Single-Dose Pharmacokinetics of Nicotine 4 mg Sublingual Tablets Versus Nicorette Lozenge 4 mg in Healthy Smokers Under Fasted Conditions
Brief Title: Pharmacokinetics of Nicotine Sublingual Tablets Versus Nicorette Lozenge in Healthy Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Rose Research Center, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16-07-239
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Use Disorder; Cigarette Smoking
Keywords: pharmacokinetics; nicotine absorption
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Administration, Sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual tablet 4 mg (Experimental): The 24 study participants will be administered the sublingual 4 mg nicotine tablet on one occasion. Blood samples will be obtained for 4 hours for analysis of nicotine plasma levels.
  Interventions: Drug: Sublingual tablet 4 mg versus Nicorette Lozenge 4mg
- Nicorette lozenge 4 mg (Active Comparator): The 24 study participants will be administered the Nicorette lozenge containing 4 mg of nicotine on one occasion. Blood samples will be obtained for 4 hours for analysis of nicotine plasma levels.
  Interventions: Drug: Sublingual tablet 4 mg versus Nicorette Lozenge 4mg

INTERVENTIONS:
Drug: Sublingual tablet 4 mg versus Nicorette Lozenge 4mg — * One dose of study drug (sublingual tablet or Nicorette Lozenge) will be administered to each subject in the morning on Day 1.
  * The second administration of drug will occur at least 48 hours after the initial administration. Subjects will receive the other dosage form and be instructed according to whether they are receiving the sublingual tablet or the lozenge.
  Other Names: Pharmacokinetic comparison of two nicotine dosage forms

SUMMARY:
The purpose of the study is to compare two different dosage forms from which nicotine is released and absorbed into the bloodstream.

DETAILED DESCRIPTION:
Objective The primary objective of this study is to determine the pharmacokinetic profile of a single dose of Nicotine Sublingual Tablets, 4 mg (Test Product) versus Nicorette Lozenge 4 mg in healthy adult smokers when administered under fasted conditions.

Study Design This is an open-label, pseudorandomized, two-way crossover comparison of the 4 mg sublingual nicotine tablet versus the Nicorette Lozenge 4 mg.

Number of Subjects Twenty-four (24) healthy adult smokers will be enrolled. Screening Procedures Demographic data, medical and medication histories, physical examination, measurement of height and weight, electrocardiogram (ECG), vital signs (blood pressure, heart rate, body temperature and respiratory rate), hematology, chemistry, urinalysis, end-expired Carbon Monoxide, and serum pregnancy test (for female subjects only) .

Confinements Subjects will be confined approximately 2 hours or earlier prior to study drug administration until after discharge vital signs and the 240 minute (min) post-dose blood draw and End-of-Study (EOS) procedures.

Study Drug Administration A single dose of Test Product (Nicotine Sublingual Tablets, 4 mg) and Nicorette Lozenge 4 mg will be administered to each subject in the study.

Sample Collection A total of 14 blood samples will be obtained per period. Samples will be taken pre-dose (up to 90 minutes prior to dose) and 3, 6, 9, 12, 15, 20 30, 45, 60, 90, 120, 180 and 240 minutes post-dose. A minimum of 48 hours will transpire between dose administrations.

Safety Assessments Vital signs (blood pressure, heart rate, body temperature and respiratory rate) will be measured before administration of study drug. The following will be performed at check-in: urine pregnancy test (for female subjects only). Ongoing monitoring for adverse events (AEs) will be performed during the study. Prior to release from the clinic, a well-being assessment and discharge vital signs will be completed 240 minutes (±60 min) post dosing or at Early Termination (ET).

End of Study (EOS) or Early Termination (ET) Procedures Vital signs and monitoring for AEs will be done 240 min post-dosing or at ET/withdrawal prior to release from clinic.

Analytical Method Plasma concentrations of nicotine will be determined using a validated liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) method.

Pharmacokinetics/Pharmacodynamics Determination of primary parameters Area under the curve ( AUC0-t, AUC0-inf), concentration maximum (Cmax), Time to maximum concentration(Tmax) and secondary parameters such as plasma elimination half-life( t1/2) using a by non-linear kinetics program (WinNonlin®). Pharmacodynamics effects will be measured by taking the heart rate and blood pressure will be taken three times in the first 30 minutes after test product administration. A craving assessment will be obtained at 1, 3, 7, 11, and 14 minutes post-medication administration.

Statistical Analyses No formal statistical analyses are planned; descriptive statistics of the concentration and pharmacokinetic data on nicotine will be provided. Exploratory analyses of craving reductions will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have to be 18-45 years old
2. Participants must provide written informed consent prior to any study related procedures being performed.
3. Participants must have a willingness and ability to comply with the protocol requirements.
4. Participants must be in good health and free from any clinically significant pathology (gastrointestinal tract, hepatic, renal, cardiovascular, CNS diseases)
5. Female participants of childbearing potential, in addition to having a negative urine pregnancy test, must be willing to use a form of birth control during the study. The hormonal contraceptives should be avoided within 2 month prior to study entry.
6. Participants must consume more than 10 cigarettes daily and Fagerström Test for Nicotine Dependence score of 4 or greater.
7. Participants must have no intention of quitting smoking in the next 60 days.

Exclusion Criteria:

1. Volunteers that have used other nicotine delivery system such as nicotine lozenge, nicotine patch, nicotine inhaler, or nicotine nasal spray etc within 30 days of study entry.
2. Volunteers who have currently involved in another clinical trial or have used any investigational drug within 3 month of study entry.
3. Volunteers who are pregnant or lactating, or plan to become pregnant within 6 months.
4. Volunteers who have diagnosed heart disease or are being treated with medication or had an irregular heartbeat or have had a myocardial infarction.
5. Volunteers with diagnosed stomach ulcers.
6. Volunteers who are taking insulin for diabetes.
7. Volunteers with high blood pressure not controlled by medication or a blood pressure greater than 150 mmHg systolic or 90 mmHg diastolic.
8. Volunteers who are unable to fulfill the visit schedule
9. Volunteers who have severe allergic history
10. Volunteers who have known intolerance to medication
11. Volunteers who have diagnosed chronic diseases of cardiovascular, pulmonary, neuro-endocrine systems, gastrointestinal, hepatic, renal, and blood diseases
12. Volunteers who had surgical operations on gastrointestinal tract with the exception of appendectomy
13. Volunteers who donated 450 mL and more of his/her blood or blood plasma within the last 2 months prior to the study entry
14. Volunteers who meet criteria for dependence on a substance other than nicotine.
15. Participants having a body mass index below 18 or over 35.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
the time course profile of nicotine absorption from the two nicotine dosage forms. | Fourteen blood samples will be collected over a 240 minute period after drug administration.

SECONDARY OUTCOMES:
Assessment of craving for a cigarette | The craving assessment will be obtained at 1, 3, 7, 11,and 14 minutes after drug administration
  Five questions about desire to smoke will be assessed using visual analog scales at the time points above.
Safety assessments: Vital signs | Vital signs will be measured prior to drug administration, 3 times in the first 30 minutes, and prior to discharge at 240 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Vocci, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Rose Research Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data may be shared with investigators who send the PI a data analysis plan.